CLINICAL TRIAL: NCT03687645
Title: 13C- Pyruvate DNP Hyperpolarised Magnetic Resonance Imaging Metabolic Assessment of Disease
Brief Title: Hyperpolarised 13C-Pyruvate MRI Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Principal Investigator, Shonit Punwani, Principal Investigator, University College, London
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 205839
Record Dates: First submitted 2018-09-11; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Cancer; Cardiovascular Diseases
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prostate Cancer (Experimental): Patients with biopsy-proven prostate cancer will be recruited for an additional Hyperpolarised MRI scan prior to any treatment
  Interventions: Diagnostic Test: Hyperpolarised MRI
- Renal Cancer (Experimental): Patients with biopsy-proven renal cell carcinoma will be recruited for an additional Hyperpolarised MRI scan prior to any treatment
  Interventions: Diagnostic Test: Hyperpolarised MRI
- Breast Cancer (Experimental): Patients with biopsy-proven breast cancer will be recruited for an additional Hyperpolarised MRI scan prior to any treatment
  Interventions: Diagnostic Test: Hyperpolarised MRI
- Lymphoma (Experimental): Patients with biopsy-proven lymphoma will be recruited for an additional Hyperpolarised MRI scan prior to any treatment
  Interventions: Diagnostic Test: Hyperpolarised MRI

INTERVENTIONS:
Diagnostic Test: Hyperpolarised MRI — Hyperpolarized (HP) 13C MR is an advanced imaging technique that allows monitoring of dynamic metabolic processes non-invasively. Hyperpolarisation is a process that provides dramatic gains in sensitivity (>10,000) of MRI signal collected from 13C-labelled substrates that can be injected into living systems, allowing in-vivo metabolism for the first time to be observed in real-time using imaging.

SUMMARY:
Metabolic changes related to disease are the precursor to anatomical changes in tissues. Currently the imaging methods routinely used in clinical practice look at the anatomical changes. Whilst these methods are very helpful in making clinical decisions, they are far from being perfect. Early disease can be missed because these methods are not sensitive enough and it is not clear whether disease is present or not. Additionally, it is also difficult to know whether disease it aggressive or non-aggressive.

Hyperpolarised MRI is a new imaging tool that may allow addressing these deficiencies in current imaging technology. The process of hyperpolarisation allows the production of an injectable solution that can produce signal on a standard MRI scanner inferring information about the metabolism occurring at a particular location. This technology has only just become available for clinical use.

The initial stages of evaluation require the investigators to refine and develop the new imaging protocols so that assessment can be made as to whether consistent results can be achieved. Additionally, refining the imaging protocol could also aid in identifying where the best potential future clinical use of this technology should be targeted.

Within this application the investigators aim to try out hyperpolarised MRI in a number of different cancers and also see whether it is useful to assess cardiac metabolism. The investigators will be using 13C-labelled metabolites (for this study 13C- pyruvate) which will allow interrogation of glucose metabolism. The derangement of glucose metabolism is common to a number of disease processes.

DETAILED DESCRIPTION:
The main objectives of this work are to generate proof-of-concept first-in-human metabolic imaging data using hyperpolarised MRI for patients with prostate cancer (n=15), renal (n=5), breast cancer (n=5), lymphoma (n=5) and cardiac diseases (n=5). Each cohort will provide sufficient value for high-impact publication and the essential preliminary data for subsequent individual grant applications. The findings will be correlated with conventional imaging and with clinical patient details and where applicable patient outcome. The study will take 3 years.

The main ethical, legal and management issues from the study are;

1. Hyperpolarised Injectable The investigators will be using a product to inject into patients that will be manufactured on site. This will be a GMP facility to ensure sterility. The methodology to do this is new. The investigators will have established safety through evaluation of the processes within the facility with institutional approval prior to utilisation of the product in patients. In addition, any product that is to be injected will be taken through a quality control module which will determine its pH, temperature, concentration and provided these are within specified safe parameters will allow the investigators to inject into the patient. The QC module itself will be validated/qualified prior to its use. Finally, solution produced for injection will go through a sterile filter and also be sent for culture. Patients will be monitored throughout the study and will be followed up after examination.
2. MRI Safety

   1. The investigators will be using new MRI coils that allows transmission of radiofrequency signals into the body and collect them. A new coil is required because the investigators need them to be tuned to the frequency of 13C (usually MRI uses 1H).
   2. The investigators will be using new MRI software that has been programmed in house to generate the signals. This software has undergone in-house and institutional approval processes to confirm that it is safe for human use.
3. Recruitment An information leaflet be dispatched to the volunteer and subsequent contact will be made to assess interest in participation and discuss arrangement for the study.

35 patients will be recruited in the first instance in one of the following ways: A. Through identification at the relevant multidisciplinary team meeting (MDT) B. Patients with confirmed cancer or heart conditions who are attending for a clinical MRI scan (or from an imaging list) as part of standard care at UCLH.

C. Direct referral from clinical colleagues D. Cancer or cardiology in-patients who are well enough and meet the recruitment criteria

Only 25/35 patients will be injected with the hyperpolarised solution. The remaining 10/35 (prostate cancer patients) will allow the investigators to optimise the MRI clinical scan technique and use of an endorectal MRI coil (to be inserted into the back passage). This optimisation will ensure that when patients with prostate cancer are evaluated with the hyperpolarised injectable, the best chance of detecting the hyperpolarised MR signal is provided.

(4) Consent Patients will have had information > 24hours in advance of consenting to study and having the research MRI. Consent will be obtained by a member of the research team trained in taking consent. Interpretation services will be made available if the patient is not fluent in spoken or written English.

(5) Data Management

1. Unexpected Findings: Any unexpected findings in participants with known cancer (e.g. unknown metastatic disease) will be directly communicated to the clinical team.
2. Confidentiality of Data: All data will be collated by the chief investigator and research team. Electronic data and images will be held on password protected databases and will be pseudo anonymised to avoid identification of patients. Adherence will be made to the data protection act 1998. Patient data will never leave UCLH. This system is compliant with UCLH data protection regulations.

   (6) Patient Burden/Benefit Patients will need to attend the hospital for the additional scan required for this study. The total amount of time that they will spend within the study is approx. 4 hours (including consent, preparation and monitoring). Patients will reimbursed for transport costs to enable them to attend for their scan.

   The investigators will where possible try to coincide the scan with a clinical appointment to minimise repeated attendances to hospital. There will be no direct benefit to patients of having undergone this scan. However, participants will contribute towards potential societal benefit if the technique is successful. The investigators will keep the doctors of the patients informed with the study results which can then be communicated to participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or over
2. Suspected Prostate Cancer/Renal Cancer/Rectal Cancer/Pancreatic Cancer
3. No current renal impairment or an eGFR within a standard reference value if there is a history of renal disease.
4. Subject able to comply with study procedures and provide informed consent.
5. Patient is willing to undergo MRI/Hyperpolarised 13C-Pyruvate MRI or with other nuclei and substrate (where appropriate).
6. Eastern Cooperative Oncology Group Performance Status (ECOG) of 0 or 2

Exclusion Criteria:

1. Contraindication to MRI (e.g cardiac pacemaker)
2. Contraindication to MR contrast agents
3. Pregnancy
4. Breast Feeding
5. Deranged renal function (eGFR<30) -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Pyruvate to Lactate conversion following the injection of Hyperpolarised 13C- Pyruvate | 3 years
  Following the injection of Hyperpolarised 13C- Pyruvate, the rate of conversion of pyruvate to lactate will be measured using the lactate spectral peak height to produce metabolic map. Such metabolic maps generate the first-in-human images of tumour metabolism in patients with prostate, renal, breast, lymphoma cancers and cardiac disease

SECONDARY OUTCOMES:
Pyruvate to Lactate conversion as an imaging biomarker | 3 years
  Pyruvate to lactate conversion rate has the potential to be used as an imaging biomarker.
  The higher rate of conversion within a tumour could be used to risk stratify the disease and as a prognostic tool.
Correlation of Hyperpolarised 13C- Pyruvate MRI with genetic markers | 3 years
  Hyperpolarised 13C- Pyruvate MRI results and pyruvate to lactate conversion rate is going to be correlated with genetic markers of disease aggressiveness to investigate whether there is any creation between the two.
  The genetic data for this analysis will be used when collected as part of routine clinical care
Hyperpolarised 13C MRI as an imaging biomarker to assess response | 3 years
  Using Hyperpolarised 13C - Pyruvate MRI, the changes in pyruvate to lactate conversion rate following chemotherapy, radiotherapy, surgery and ablative technique will be assessed.
  These changes will then be correlated with clinical outcome measures that are routinely used in patients' managements to investigate the potential of hyperpolarised 13C - Pyruvate MRI for response monitoring in different cancer subtypes.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shonit Punwani, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No